CLINICAL TRIAL: NCT01992445
Title: Suicidal Thought and Biological Markers: A Prospective Multicenter Study Validating Verbal, Non-verbal and Genetic Methods to Assess Suicidal Intent
Brief Title: Suicidal Thought and Biological Markers
Acronym: STM
Status: Completed | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Other Study IDs: 20133770
Record Dates: First submitted 2013-11-08; First posted 2013-11-25 (Estimated); Last update posted 2016-05-23 (Estimated); Status verified 2016-05

CONDITIONS: Suicidal Intention
Keywords: suicide; suicidal intent; thought markers
MeSH Terms: conditions — Suicide

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Buccal swabs
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Suicidal
- Other mental health
- Control (non suicidal, non mental health)

SUMMARY:
Thought Markers (Tm) and Biomarkers(Bm) to accurately predict the likelihood of a repeated suicide attempt.

DETAILED DESCRIPTION:
The purpose of this study is to develop a predictive model that includes Thought Markers (Tm) and Biomarkers(Bm) to accurately predict the likelihood of a repeated suicide attempt.

ELIGIBILITY:
Inclusion Criteria:

oBe able to understand the requirements of the study and provide written informed consent to participate in this study. Signed and dated informed consent will be obtained from each patient before participation in the study, oHave provided written authorization for the use and disclosure of their protected health information, oBe 13 years of age or older, oBe diagnosed with: oSuicide ideation/attempts/gestures, or oNon-suicidal and having other mental disorders, oNon-mentally ill, and non-suicidal controls, oSpeak English as the primary language in the home, oAgree to abide by the study protocol and its restrictions and be able to complete all aspects of the study.

Exclusion Criteria:

oSignificant unstable medical condition that may obscure the scientific interpretability of the study or unduly increase the risks of the protocol, oAnticipated inability to attend follow-up phone interview, oPatients whose level of consciousness precludes consent and research assessments, oPatients unable to assent because of severe mental retardation, oPatients who in the judgment of the Investigator may be unreliable or uncooperative with the evaluation procedure outlined in this protocol, oFor control patients a diagnosis of depression or another non-mental illness, or a history of suicidal behavior or suicidal attempt, oPatients who are unwilling to provide the DNA sample.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Emergency Department and inpatients
Sampling Method: Non-Probability Sample
Enrollment: 375 (Actual)
Dates: Start 2013-10; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Columbia Suicide Severity Rating Scale | 1 month
  Questionnaire

SECONDARY OUTCOMES:
Acoustic analysis of voice | 1 month
  Voice recording
Video analysis | Baseline
  Video recording
DNA analysis | Baseline
  DNA analysis

CONTACTS AND LOCATIONS:
Overall Officials: John Pestian, PhD, Study Director — CCHMC
Locations (3):
- United States (3):
  - CCHMC, Cincinnati, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - Princeton Community Hospital, Princeton, West Virginia